CLINICAL TRIAL: NCT07220824
Title: GUselkumab for the Treatment of PsA: Effectiveness Results by Ultrasound
Brief Title: A Study of Guselkumab in Participants With Psoriatic Arthritis (PsA) in a Real-World Setting
Acronym: GURU
Status: Recruiting | Type: Observational
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: CNTO1959PSA4020; CNTO1959PSA4020 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2025-10-22; First posted 2025-10-24 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Arthritis, Psoriatic
MeSH Terms: conditions — Arthritis, Psoriatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Group 1: Psoriatic Arthritis: Participants with confirmed diagnosis of psoriatic arthritis treated with guselkumab as per standard clinical practice will be enrolled. No drug will be provided as part of this study. Only data available within routine clinical practice, including results of ultrasound examinations, will be collected in this study. Additionally, questions will be asked from participants about their health and well-being.

SUMMARY:
The purpose of this study is to assess how well guselkumab works in improving symptoms of psoriatic arthritis (an inflammatory disease that affects the joints in participants with psoriasis, a skin condition that causes red, scaly patches) using muscoloskeletal ultrasound (MSUS) in a real-world setting.

ELIGIBILITY:
Inclusion criteria:

* Diagnosis of PsA as per CASPAR classification criteria for at least six months with active PsA defined as a tender joint count (TJC) greater than or equal to (>=) 3/68 and a swollen joint count (SJC) >= 3/66 at baseline, or C-reactive protein (CRP) >=0.3 milligrams per deciliter (mg/dL) if TJC and/or SJC are less than (<) 3
* a) Total synovitis power doppler ultrasound (PDUS) score >=2 and inflammation related to power doppler (PD) signal >=2 for at least 1 affected joint of 48 joints at the baseline visit (before first Guselkumab administration), or b) Total synovitis PDUS score >=2 and inflammation related to PD signal >=1 for at least 2 affected joints of 48 joints at the baseline visit (before first Guselkumab administration)
* Start guselkumab for the indication of PsA as part of standard clinical practice at the time of enrollment into the observational study or within a maximum of two weeks after the initial baseline visit
* Participants must be biologic-naïve or previously exposed to only one biologic Disease-Modifying Antirheumatic Drugs (bDMARD) and/or apremilast/deucravacitinib
* At least one clinically involved enthesitis site, defined by SPARCC index >= 1, and one imaging-detected enthesitis site at baseline

Exclusion criteria:

* Previous exposure to Guselkumab or to more than one bDMARD for any indications
* Prior treatment with Janus kinase (JAK) inhibitors
* Contraindications to Guselkumab as per the summary of product characteristics (SmPC)
* Current enrollment in other investigational study or participation in other investigational study completed from less than 30 days
* Current enrollment in an observational study with Guselkumab sponsored or managed by sponsor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will include participants affected with PsA according to classification for psoriatic arthritis (CASPAR) criteria.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-12-04 (Actual); Primary Completion 2027-07-31 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Percentage Reduction From Baseline in Global OMERACT and EULAR Synovitis Score (GLOESS) at Week 12 | Baseline and Week 12
  GLOESS is an ultrasound scoring system to assess the presence and severity of synovitis measured for 24 pairs of joints. The scoring is from 0 to 3 for each joint where 0: No abnormalities or changes, 1: Mild changes, 2: Moderate changes and 3: Severe changes. The total score for 48 joints can range from 0 to 144, where higher score indicates more inflammation.
Percentage of Participants Achieving Disease Activity Index for Psoriatic Arthritis (DAPSA) Low Disease Activity (LDA) Score Less Than or Equal to 14, at Week 24 | Week 24
  Percentage of participants achieving DAPSA LDA (that is, a score less than or equal to [<=] 14) will be reported. DAPSA assesses the joint domain of PsA and is derived from the sum of the following components: Participant's assessment of pain on visual analog scale (VAS ; 0-10 centimeters [cm]; VAS 0= excellent; 10= poor), Participant's global assessment of disease activity on VAS (0 to 10 cm VAS, 0=excellent and 10=poor), tender joint count (0-68), swollen joint count (0-66) and C-reactive protein (CRP) level. A higher score indicates more active disease activity.

SECONDARY OUTCOMES:
Percentage of Participants Achieving Resolution of Enthesitis by Ultrasound at Week 12 | Week 12
  Enthesitis is assessed by ultrasound using the Global Outcome Measures in Rheumatology (OMERACT) enthesitis score which scores 6 pairs of entheses bilaterally: common extensor tendon, quadriceps tendon, patellar tendon at proximal and distal insertion, achilles tendon and plantar aponeurosis. Each affected entheses out of the 6 bilateral sites will be scored according to OMERACT enthesitis composite semiquantitative scale (range 0-3) and the sum of each single abnormal site of the 6 bilateral targeted entheses is represented by Global OMERACT score ranging from 0-48. A higher score indicates more active disease activity.
Percentage Reduction from Baseline in Spondyloarthritis Research Consortium of Canada (SPAARC) Index at Week 24 | Baseline and Week 24
  The SPARCC developed a measure for enthesitis in general spondyloarthritis which focuses on the clinical evaluation and validation of the following 16 entheseal sites: greater trochanter (Right/Left); quadriceps tendon insertion into the patella (Right/Left); patellar ligament insertion into the patella and tibial tuberosity (Right/Left); achilles tendon insertion (Right/Left); plantar fascia insertion (Right/Left); medial epicondyles (Right/Left); lateral epicondyles (Right/Left); supraspinatus insertion (Right/Left). Each entheseal site is assessed for tenderness on a dichotomous basis, i.e., 0= non-tender, 1= tender, for a total score ranging from 0 to 16. Higher scores indicate more severe enthesitis. Negative changes from baseline indicate improvement of enthesitis.
Percentage of Participants Achieving DAPSA Remission at Week 24 | Week 24
  DAPSA assesses the joint domain of PsA where a higher score indicates more active disease activity. DAPSA remission indicates DAPSA score of 4 or less. DAPSA remission signifies a greater reduction in disease activity, with minimal or no symptoms when compared with DAPSA LDA.
Percentage of Participants Achieving DAPSA LDA/Remission at Week 52 | Week 52
  DAPSA assesses the joint domain of PsA where a higher score indicates more active disease activity. DAPSA remission indicates DAPSA score of 4 or less. DAPSA LDA indicates DAPSA score of 14 or less. DAPSA remission signifies a greater reduction in disease activity, with minimal or no symptoms when compared with DAPSA LDA.
Number of Participants Achieving Minimal Disease Activity (MDA) at Weeks 12, 24 and 52 | At Weeks 12, 24 and 52
  MDA status is defined by meeting 5 of 7 criteria: tender joint count <= 1; swollen joint count <=1; psoriasis area and severity index (PASI) <=1 or body surface area (BSA) with PsO <=3 percent (%); participant's VAS pain score of <=15; participant's VAS global disease activity score of <=20; disability index of the health assessment questionnaire (HAQ-DI) score <=0.5; and tender entheseal points <=1.
Percentage of Participants Achieving Reduction in VAS Pain Scores at Week 12 and 24 | At Weeks 12, and 24
  The pain VAS is a self-administered assessment of average pain during the past week. The scale ranges from "no pain" (0 mm) to "the worst possible pain" (100 mm). Higher scores indicate more pain.
Number of Participants with Improvement in Health Assessment Questionnaire Disability Index (HAQ-DI) At Weeks 12 and 24 | At Weeks 12 and 24
  HAQ-DI is used to assess the long-term influence of chronic disease on a participant's level of functional ability and activity restriction. The HAQ-DI includes questions of fine movements of the upper extremity, locomotor activities of the lower extremity, and activities that involve both upper and lower extremities. For each question the score is from 0 (without any difficulty) to 3 (unable to do) where lower scores are indicative of better functioning and higher score reflects worse function.
Number of Participants with Persistence to Guselkumab Treatment up to 52 Weeks | Up to Week 52
  Number of participants who were persistent with guselkumab treatment up to 52 weeks after initiation will be reported.
Number of Participants with Adverse Events (AEs) | Up to Week 52
  An AE is any untoward medical occurrence in a participating patient administered a medicinal product. An AE does not necessarily have a causal relationship with the treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (15):
- Italy (15):
  - Policlinico di Bari, Bari
  - Hospital Carlo Urbani, Iesi
  - IRCCS Ospedale Galeazzi Sant Ambrogio, Milan
  - Istituto Ortopedico Gaetano Pini, Milan
  - San Raffaele Hospital, Milan
  - ASST Grande Ospedale Metropolitano Niguarda, Milan
  - Azienda Ospedaliera Universitaria Federico II, Napoli
  - Azienda Ospedaliero Universitaria Policlinico Paolo Giaccone, Palermo
  - Fondazione IRCCS Policlinico San Matteo, Pavia
  - Ospedale Santa Chiara AO Universitaria Pisana, Pisa
  - Arcispedale Santa Maria Nuova - IRCCS, Reggio Emilia
  - Fondazione Policlinico Universitario A Gemelli IRCCS, Roma
  - A O Universitaria Senese Ospedale Santa Maria alle Scotte, Siena
  - AO Ordine Mauriziano, Torino
  - Azienda Ospedaliera Universitaria Integrata Verona, Verona

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of Johnson & Johnson Innovative Medicine is available at www.innovativemedicine.jnj.com/our-innovation/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu.
URL: https://innovativemedicine.jnj.com/our-innovation/clinical-trials/transparency